CLINICAL TRIAL: NCT03248076
Title: Effect of Fentanyl on Expression of Main Opioid Receptor (OPRM1) on Human Granulosa Cells During Ultrasound-guided Transvaginal Oocyte Retrieval.
Brief Title: Effect of Fentanyl on Main Opioid Receptor (OPRM1) on Human Granulosa Cells.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: George Papanicolaou Hospital (Other)
Collaborators: Papanikolaou Evaggelos (Unknown); Naidecki Robert (Unknown); Pakaki Fay (Unknown); Raikos Nikolaos (Unknown)
Responsible Party: Principal Investigator, Asouhidou Irene, Assisting Professor, George Papanicolaou Hospital
Other Study IDs: Opioids-OPU
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Stress Reaction; Opioid Use
MeSH Terms: conditions — Fractures, Stress | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fentanyl citrate: Baseline blood sample and oocyte fluid will be collected under propofol anesthesia. Fifteen minutes after administration of 1γ/kgfentanyl, it will be collected again blood sample and oocyte fluid. Cortisone and fentanyl level will be measured in all samples.
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl Citrate — 1γ/Kg fentanyl

SUMMARY:
Opioids is known that produce not only analgesia but also hyperalgesia through activation of central glutaminergic system-GABA. At the same time, recently it was found that the main opioid receptor (OPRM1) is present on human granulosa cells and exogenous opiates and their antagonists can influence granulosa cell vascular endothelial growth factor (VEGF) production via OPRM1, causing ovarian hyperstimulation syndrome.

This study aims to investigate if a single exposure to opioids is enough to produce activation of stress mechanism during oocyte retrieval.

DETAILED DESCRIPTION:
The main opioid receptor (OPRM1) is present on human granulosa cells and exogenous opiates and their antagonists can influence granulosa cell vascular endothelial growth factor (VEGF) production via OPRM1, causing ovarian hyperstimulation syndrome.

This study aims to investigate if a single exposure to opioids is enough to produce activation of stress mechanism during ultrasound-guided oocyte retrieval. It will be measured the level of cortisone before and 15min after iv administration of fentanyl on blood and on oocyte fluid.

ELIGIBILITY:
Inclusion Criteria:

* American Physical Status I-III, BMI<30,

Exclusion Criteria:

* Heart failure
* hepatic failure, hepatitis,
* drug abuse
* receiving b blockers
* receiving b agonists (even bronchodilators)

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers oocyte donor
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-10-10 (Estimated)

PRIMARY OUTCOMES:
fentanyl | 15 minutes
  fentanyl on blood sample and oocyte fluid

SECONDARY OUTCOMES:
cortisone | 15 min
  cortisone on blood sample and oocyte fluid

CONTACTS AND LOCATIONS:
Overall Officials: Irene Asouhidou, MD, PhD, Principal Investigator — Assisting Nature
Locations (1):
- Section of Anatomy, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bottcher B, Seeber B, Leyendecker G, Wildt L. Impact of the opioid system on the reproductive axis. Fertil Steril. 2017 Aug;108(2):207-213. doi: 10.1016/j.fertnstert.2017.06.009. Epub 2017 Jun 29. PMID 28669481
- [Background] Lunger F, Vehmas AP, Furnrohr BG, Sopper S, Wildt L, Seeber B. Opiate receptor blockade on human granulosa cells inhibits VEGF release. Reprod Biomed Online. 2016 Mar;32(3):316-22. doi: 10.1016/j.rbmo.2015.12.006. Epub 2016 Jan 6. PMID 26803207
- [Background] Kouvaras E, Asprodini EK, Asouchidou I, Vasilaki A, Kilindris T, Michaloudis D, Koukoutianou I, Papatheodoropoulos C, Kostopoulos G. Fentanyl treatment reduces GABAergic inhibition in the CA1 area of the hippocampus 24 h after acute exposure to the drug. Neuropharmacology. 2008 Dec;55(7):1172-82. doi: 10.1016/j.neuropharm.2008.07.025. Epub 2008 Jul 26. PMID 18706433